CLINICAL TRIAL: NCT01184989
Title: An Open Label, Non-comparative, Pharmacokinetic and Pharmacodynamic Study to Evaluate the Effect of Dabigatran Etexilate on Coagulation Parameters Including a Calibrated Thrombin Time Test in Patients With Moderate Renal Impairment (Creatinine Clearance 30-50 ml/Min) Undergoing Primary Unilateral Elective Total Knee or Hip Replacement Surgery
Brief Title: Treatment of Patients Undergoing Primary Unilateral Elective Total Knee or Hip Replacement With Dabigatran Etexilate
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 1160.86; 2010-018723-26 (EudraCT Number: EudraCT)
Record Dates: First submitted 2010-08-16; First posted 2010-08-19 (Estimated); Results first posted 2014-05-23 (Estimated); Last update posted 2018-09-25 (Actual); Status verified 2018-08

CONDITIONS: Arthroplasty, Replacement; Prevention of Venous Thromboembolism; Moderate Renal Impairment (CrCl 30-50 mL/Min)
MeSH Terms: interventions — Dabigatran

ARMS (1):
- Dabigatran etexilate (Other): open label, once daily dose approved by EMEA and Health Canada
  Interventions: Drug: Dabigatran etexilate

INTERVENTIONS:
Drug: Dabigatran etexilate — once daily approved dose by EMEA and Health Canada

SUMMARY:
To supplement the current evidence of the effect of Pradaxa® (dabigatran etexilate) on coagulation parameters, including a calibrated thrombin time test, in patients with moderate renal impairment undergoing elective total hip- or knee-replacement surgery, this PK/PD study will be conducted.

ELIGIBILITY:
Inclusion criteria:

1. Patients scheduled for primary unilateral elective total knee or hip replacement, male or female being 18 years or older
2. Moderate renal impairment (CrCl 30-50 mL/min)
3. Written informed consent
4. Caucasian patients

Exclusion criteria:

1. Patients weighing less than 40 kg.
2. Patients requiring chronic treatment with anticoagulants (e.g. vitamin K antagonists; e.g. patients with atrial fibrillation, patients with artificial heart valves, etc.).
3. Patients who in the investigator's judgment were perceived as having an excessive risk of bleeding, for example:

   Constitutional or acquired coagulation disorders

   History of bleeding diathesis

   Clinically relevant bleeding (gastrointestinal, pulmonary, intraocular or urogenital bleeding) within 3 months of enrolment

   Major surgery or trauma (e.g. hip fracture) within 3 months of enrolment

   History of thrombocytopenia, including heparin-induced thrombocytopenia, or a platelet count <100 000 cells/microliter at randomization

   Any history of hemorrhagic stroke or any of the following intracranial pathologies: bleeding, neoplasm

   Any arteriovenous malformations, vascular aneurysms or major intraspinal or intracerebral vascular abnormalities

   Presence of malignant neoplasms at higher risk of bleeding

   Known or suspected oesophageal varices

   Symptomatic or endoscopically documented gastroduodenal ulcer disease in the previous 30 days

   Treatment with anticoagulants, clopidogrel, ticlopidine, abciximab, aspirin >162.5 mg/day or non-steroidal anti-inflammatory drug (NSAID) with t1/2>12 hours within 7 days prior to hip or knee replacement surgery OR anticipated need while the patient was receiving study medication and prior to 24 hours after the last administration of study medication (COX-2 selective inhibitors are allowed) because of anticipated need of quinidine, verapamil or other restricted medication during the treatment period
4. Recent unstable cardiovascular disease (in the investigator's opinion) such as uncontrolled hypertension, that was ongoing at the time of enrolment or history of myocardial infarction within 3 months of enrolment.
5. Ongoing treatment for VTE.
6. Liver disease expected to have any potential impact on survival (i.e. hepatitis B or C, cirrhosis) or ALT/AST >3x upper limit of normal range (ULN). This did not include Gilbert's syndrome or hepatitis A with complete recovery.
7. Known severe renal insufficiency (CrCl <30 mL/min) and patients with mild renal insufficiency (CrCl >50 mL/min) or normal renal function.
8. Planned anaesthesia with post-operative indwelling epidural catheters.
9. Pre-menopausal women (last menstruation <=1 year prior to signing informed consent), who were:

   Pregnant

   Nursing

   Of child-bearing potential and were NOT practicing acceptable methods of birth control, or did NOT plan to continue practicing an acceptable method throughout the study. Acceptable methods of birth control included intrauterine device; oral, implantable or injectable contraceptives and surgical sterility
10. Hypersensitivity to dabigatran etexilate or to any of excipients.
11. Participation in a clinical trial within 30 days of enrolment.
12. Known alcohol or drug abuse which would interfere with completion of the study; patients considered unreliable by the investigator concerning the requirements for follow-up during the study and/or compliance with study drug administration.
13. Previous participation in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 142 (Actual)
Dates: Start 2010-08; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (10):
- Austria (2):
  - 1160.86.43001 Boehringer Ingelheim Investigational Site, Graz
  - 1160.86.43003 Boehringer Ingelheim Investigational Site, Vienna
- Canada (3):
  - 1160.86.01001 Boehringer Ingelheim Investigational Site, Red Deer, Alberta
  - 1160.86.01002 Boehringer Ingelheim Investigational Site, Halifax, Nova Scotia
  - 1160.86.01003 Boehringer Ingelheim Investigational Site, Charlottetown, Prince Edward Island
- 1160.86.42002 Boehringer Ingelheim Investigational Site, Prague, Czechia
- 1160.86.35801 Boehringer Ingelheim Investigational Site, Jyväskylä, Finland
- 1160.86.31002 Boehringer Ingelheim Investigational Site, Hilversum, Netherlands
- Sweden (2):
  - 1160.86.46002 Boehringer Ingelheim Investigational Site, Hässleholm
  - 1160.86.46001 Boehringer Ingelheim Investigational Site, Mölndal

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 30 patients did not receive any study medication.
Groups:
- Patients Treated With Dabigatran Etexilate: Patients treated with Dabigatran Etexilate 150mg once daily. At the day of surgery the treatment will be initiated 1-4 h post surgery with 75mg.
  142 patients were enrolled for the study, but only 112 were treated. Therefore, the number of started patients corresponds to the ones that were actually treated.
Period: Overall Study
Arm/Group | Patients Treated With Dabigatran Etexilate
Started | 112 (Treated Patients)
Completed | 100
Not Completed | 12
Not completed — Adverse Event | 11
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Population: Treated Set (TS): Patients who were dispensed study medication and were documented to have taken at least one dose of investigational treatment.
Groups:
- Patients Treated With Dabigatran Etexilate: Patients treated with Dabigatran Etexilate 150mg once daily. At the day of surgery the treatment will be initiated 1-4 h post surgery with 75mg.
Arm/Group | Patients Treated With Dabigatran Etexilate
Number analyzed (Participants) | 112
Age, Continuous [Mean (Standard Deviation); unit: years] | 79.1 (6.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 78
  Male | 34

OUTCOME MEASURES:

1. Primary Outcome: Dabigatran Concentration in Plasma, Estimated From Local Hemoclot®
Description: The Hemoclot® test kit measures the dTT (diluted Thrombin time). In the present trial, as a first step, the dTT in calibration samples that had known Dabigatran concentrations was measured locally with the Hemoclot® test kit, and a linear calibration curve was fitted to the data from the calibration samples. Thereafter, for each patient at each time-point, the dTT was measured with the Hemoclot® kit and the Dabigatran concentration was read off from the calibration curve.
  These estimated concentrations are compared with concentrations measured in parallel with HPLC-MS/MS.
  As the trial objective is the method comparison and not the detection of the absolute concentrations of either of the methods, the result is reported as a relative bioavailability [%], see "Statistical Analysis 1" below. Only concentrations >= LLOQ (Lower Limit of concentration) are included in the quantitative comparison.
Time Frame: Screening, day of surgery 1 hour (h) and 2h after drug intake (di) for late finalization of surgery, 4h and 8h after di for early finalization of surgery, 15 minutes (min) before di at days 2, 3, 4, 5 and 6, at day 6 also 1h, 2h, 4h, 8h and 24 after di
Population: Correct calculation set: all patients of the Per Protocol set (PPS) (patients with at least one pair of observations for both PD and PK parameters without important protocol violations) and additionally all patients of the TS whom the only reason for not being in the PPS was the non-influential forbidden concomitant medication or vomiting
Measure: Number; unit: measurements estimated as above LLOQ
Units Other Than Participants: Measurements
Arm/Group | Patients Treated With Dabigatran Etexilate
Number analyzed (Participants) | 99
Number analyzed (Measurements) | 320
measurements estimated as above LLOQ | 136 (NA)
Statistical Analysis 1: Comparison: Patients Treated With Dabigatran Etexilate; Estimated local measurements are compared to HPLC-MS/MS measurements. The comparison was done for the 136 quantifiable measurements; Test type: Non-Inferiority or Equivalence — Bioavailability analysis; Geometric Mean; Ratio = 102.16, 90% CI [97.640 to 106.893], Standard Deviation 22.8 — Dispersion value is actually the intraindividual gCV

2. Primary Outcome: Dabigatran Concentration in Plasma, Estimated From Central Hemoclot®
Description: The Hemoclot® test kit measures the dTT (diluted Thrombin time). In the present trial, as a first step, the dTT in calibration samples that had known Dabigatran concentrations was measured centrally with the Hemoclot® test kit, and a linear calibration curve was fitted to the data from the calibration samples. Thereafter, for each patient at each time-point, the dTT was measured with the Hemoclot® kit and the Dabigatran concentration was read off from the calibration curve.
  These estimated concentrations are compared with concentrations measured in parallel with HPLC-MS/MS.
  As the trial objective is the method comparison and not the detection of the absolute concentrations of either of the methods, the result is reported as a relative bioavailability [%], see "Statistical Analysis 1" below. Only concentrations >= LLOQ (Lower Limit of concentration) are included in the quantitative comparison.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Number; unit: measurements estimated as above LLOQ
Units Other Than Participants: Measurements
Arm/Group | Patients Treated With Dabigatran Etexilate
Number analyzed (Participants) | 97
Number analyzed (Measurements) | 1158
measurements estimated as above LLOQ | 468
Statistical Analysis 1: Comparison: Patients Treated With Dabigatran Etexilate; Estimated central measurements are compared to HPLC-MS/MS measurements. The comparison was done for the 468 quantifiable measurements; Test type: Non-Inferiority or Equivalence — Bioavailability analysis; Geometric Mean; Ratio = 92.37, 90% CI [90.079 to 94.719], Standard Deviation 23.5 — The Dispersion Value is actually the intraindividual gCV

3. Primary Outcome: Dabigatran Concentration in Plasma, Measured With HPLC-MS/MS
Description: Dabigatran Concentration in Plasma, measured with HPLC-MS/MS - Most relevant timepoints are reported here, ie timepoints of day 6
Time Frame: At day 6 before drug intake (di), at 1h, 2h, 4h, 8h and 24h after di
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Patients Treated With Dabigatran Etexilate
Number analyzed (Participants) | 96
ng/mL
  before intake(N=96) | 47.5 (84.7)
  after 1h(N=93) | 87.8 (81.9)
  after 2h(N=91) | 147 (85.2)
  after 4h(N=88) | 157 (84.8)
  after 8h(N=93) | 119 (78.1)
  after 24h(N=86) | 47.7 (90.5)

ADVERSE EVENTS:
Time Frame: Up to 14 days
Arm/Group | Patients Treated With Dabigatran Etexilate
Serious Adverse Events (participants affected / at risk) | 10/112
Other Adverse Events (participants affected / at risk) | 99/112
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Patients Treated With Dabigatran Etexilate (N=112)
Gastric ulcer (Gastrointestinal disorders) | 2
Haematemesis (Gastrointestinal disorders) | 2
Gastritis haemorrhagic (Gastrointestinal disorders) | 1
Diverticulitis (Infections and infestations) | 1
Pyelonephritis (Infections and infestations) | 1
Urinary tract infection (Infections and infestations) | 1
Urosepsis (Infections and infestations) | 1
Atrial fibrillation (Cardiac disorders) | 1
Acute myocardial infarction (Cardiac disorders) | 1
Wound secretion (Injury, poisoning and procedural complications) | 1
Post procedural drainage (Surgical and medical procedures) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Patients Treated With Dabigatran Etexilate (N=112)
Anaemia (Blood and lymphatic system disorders) | 7
Dizziness (Nervous system disorders) | 14
Hypotension (Vascular disorders) | 11
Haematoma (Vascular disorders) | 6
Nausea (Gastrointestinal disorders) | 45
Vomiting (Gastrointestinal disorders) | 37
Constipation (Gastrointestinal disorders) | 11
Arthralgia (Musculoskeletal and connective tissue disorders) | 23
Urinary retention (Renal and urinary disorders) | 7
Oedema peripheral (General disorders) | 9
Pyrexia (General disorders) | 7
Haemoglobin decreased (Investigations) | 11
Wound haematoma (Injury, poisoning and procedural complications) | 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Any publication of the result of this trial must be consistent with the Boehringer Ingelheim publication policy. The rights of the investigator and of the sponsor with regard to publication of the results of this trial are described in the investigator contract.